CLINICAL TRIAL: NCT01096199
Title: A Phase I Study of TS-1, Cisplatin & RAD001 (Everolimus)
Brief Title: A Study of TS-1, Cisplatin (CDDP) and RAD001 (Everolimus)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: PK02/12/09
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Cancer
Keywords: The purpose of the study is to evaluate the safety and feasibility of combining TS-1/CDDP with RAD001. Primary; Objectives; To determine the MTD/recommended phase II dose of TS-1/CDDP/RAD001 combination -To determine; the safety of TS-1/CDDP/RAD001 combination Secondary Objectives -To preliminarily describe any clinical activity in; platinum refractory disease; To assess to effect of concurrent TS-1/CDDP on RAD001 pharmacokinetics -To explore; the relationship of tumour biomarkers and treatment response
MeSH Terms: conditions — Neoplasms | interventions — Cisplatin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TS-ONE, Cisplatin, RAD001

SUMMARY:
Hypothesis: The addition of RAD001 to TS-1/CDDP is safe and can improved the efficacy of TS-1/CDDP. The rationale for combining RAD001 with TS-1/CDDP are:

1. Potential synergism for the combination TS-1/CDDP Activation of the PI3K/AKT/mTOR pathway is frequently a characteristic of worsening prognoses (through increased aggressiveness), resistance to treatment, extension of disease and progression. The antitumour effect of RAD001 is mediated through the antiproliferative and antiangiogenic activity of mTOR inhibition. In preclinical study, RAD001 demonstrated synergism with CDDP in several cancer types including lung (A549; CI 0.47), epidermoid cancer (KB-31; CI 0.74), colon cancer (HCT116; CI 0.47) and gastric cancer (SNU 1; CI 0.204, SNU 216; CI 0.546, SNU 638; CI 0.039, SNU 668; CI 0.396) (IB, Lee 2008 AACR).
2. Potential for overcoming TS-1/CDDP resistance. Upregulation of Akt pathway was found to be an important mechanism for acquired resistance to CDDP (Lee 2005 Gyn Onc, Liu 2007 Cancer Res). In addition, gastric cancers with upregulated Akt pathway are associate with primary resistance to 5- fluorouracil, adriamycin, mitomycin C, and cisplatin (Oki 2007 PASCO)
3. Overlapping antitumour activities with TS-1/CDDP RAD001 is effective and well tolerated against subcutaneous tumours established from a variety of tumour cell lines of diverse histotypes (NSCLC, pancreatic, gastric, colon, renal, melanoma, epidermoid), including a Pgp170-overexpressing, multi-drug resistant tumor line. Partial response to single agent RAD001 was seen in a patient with gastric cancer at the dose of 5mg/day and 2 patients (gastric and oesophageal cancer) at the dose of 10mg/day, in study C2101 and C1101 respectively. A clinical benefit (stable disease, partial response and complete response) was observed in 55% of patient with gastric cancer who had failed 1st line therapy (Yamada 2009 GCS ASCO). A phase III study of RAD001 in patients with 2nd/3rd line gastric cancer has currently opened for recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented locally advanced, metastatic or recurrent solid malignancies that are refractory to standard therapy, for which convention therapy is not effective or platinum/fluoropyrimidine is indicated.
* At least one measurable or evaluable disease defined by RECIST
* Age >21 years old
* Performance status (ECOG) 0-2
* Life expectancy >3 months
* No significant problems for oral intake and drug administration
* Adequate organ functions:

  * bone marrow function (ANC ≥ 1,500/uL, Platelet ≥ 100,000/ uL, Hb ≥ 9.0 g/dl)
  * renal function: serum creatinine ≤ UNL (if serum creatinine > ULN, creatinine clearance should be ≥ 60 mL/min)
  * hepatic function (Total bilirubin < 2 x UNL and AST/ALT levels < 3 x ULN without liver metastasis, total bilirubin < 3x ULN and AST/ALT levels < 5 x ULN with liver metastasis)
* Prior systemic therapy (eg, cytotoxic chemotherapy or biologic therapy) and major surgery are allowed if at least 28 days has elapsed between completion of therapy and administration of study drugs
* Ability to understand and willingness to sign a written informed consent before study entry

Exclusion Criteria:

* Failure to recover from the reversible effects of previous chemotherapy, radiotherapy, hormonal, or biologic therapy prior to enrollment
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
* Prior radiotherapy was administered to target lesions selected for this study, or radiotherapy to the non-target lesions has been completed within 4 weeks before randomization
* Prior mTOR inhibitor
* Presence of symptomatic or progressing CNS metastasis
* Serious illness or medical conditions:

  * Congestive heart failure (NYHA class III or IV), unstable angina or myocardial infarction within the past 12 months
  * Significant arrhythmias requiring medication and conduction abnormality such as over 2nd degree AV block
  * Uncontrolled hypertension
  * Hepatic cirrhosis (≥ Child class B)
  * Interstitial pneumonia
  * Psychiatric disorder that may interfere with protocol compliance
  * Unstable diabetes mellitus
  * Uncontrolled ascites or pleural effusion
  * Active infection
  * Receiving a concomitant treatment interacting with TS-1, cisplatin or RAD001. Flucytosine (a fluorinated pyrimidine antifungal agent) Antivirals such as sorivudine, ramivudine, brivudine or other chemically related agents, warfarin, phenprocoumon, phenytoin, allopurinol, immunosuppressive agents. Strong and moderate inhibitors or inducers of P-glycoprotein, CYP3A4 and CYP3A5 (appendix A) are not eligible; a minimal of 2 weeks wash- out period will be required after stop such medications
* Known hypersensitivity to TS-1, CDDP or mTOR inhibitor.
* Pregnant or lactating woman. Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential
* Any patients judged by the investigator to be unfit to participate in the study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Liu LZ, Zhou XD, Qian G, Shi X, Fang J, Jiang BH. AKT1 amplification regulates cisplatin resistance in human lung cancer cells through the mammalian target of rapamycin/p70S6K1 pathway. Cancer Res. 2007 Jul 1;67(13):6325-32. doi: 10.1158/0008-5472.CAN-06-4261. PMID 17616691
- [Background] Lee S, Choi EJ, Jin C, Kim DH. Activation of PI3K/Akt pathway by PTEN reduction and PIK3CA mRNA amplification contributes to cisplatin resistance in an ovarian cancer cell line. Gynecol Oncol. 2005 Apr;97(1):26-34. doi: 10.1016/j.ygyno.2004.11.051. PMID 15790433